CLINICAL TRIAL: NCT04482101
Title: Single Visit Root Canal Treatment :Incidence of Postoperative Pain Using Two Different Sealers : A Randomized Clinical Trial
Brief Title: Single Visit Root Canal Treatment :Incidence of Postoperative Pain Using Two Different Sealers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Muna Abubaker Beshir Mohamed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: postoperative pain
Record Dates: First submitted 2020-07-16; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Root Canal Obturation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ah-Plus sealer (Experimental): Root canal sealer which is a resin-based formula with excellent radiopacity , low shrinkage , low solubility and outstanding flow characteristics .
  It features a 1:1 , paste-to-paste mixing system for fast , easy preparation and less waste . It is biocompatible and silver free .
  Interventions: Other: Root canal obturation
- Endosequence BC sealer (Experimental): It is a root canal sealer which is premixed ready-to-use injectable bioceramic cement paste developed for permanent root canal filling and sealing applications.
  It is insoluble , radiopaque and aluminum-free material based on calcium silicate composition , which requires the presence of water to set and hardens . It does not shrink during setting and demonstrate excellent physical properties .
  Interventions: Other: Root canal obturation

INTERVENTIONS:
Other: Root canal obturation — Root canal filling
  Other Names: Root canal sealer

SUMMARY:
The aim of this randomized clinical trial was to compare the potential effects of resin-based and bio ceramic sealers on the occurrence and intensity of postoperative pain in patients with asymptomatic apical periodontitis (AAP) .

DETAILED DESCRIPTION:
Reports about postoperative pain in endodontics range from 3%-58% in different studies .

Pain can be provoked by mechanical, chemical, or microbiological injuries to periodontal tissues . A number of treatment related parameters have been shown to be associated with the presence of postoperative pain, including working length (WL) estimation with an apex locator connected to every file , the number of visits , the choice of instrumentation , and the choice of root canal sealer .

Sealers placed in the root canals interfere with periodontal tissues through the apical foramina, lateral canals, or leaching and can potentially affect the healing process in the periodontium. Thus, the local inflammation caused by root canal obturation materials may result in postoperative pain. The intensity of inflammatory reactions depends on a number of different factors, including the composition of the sealer .

The use of a sealer during root canal obturation is essential for success of root canal treatment. The sealer has various functions:

* Attainment of impervious seal
* Filler for canal irregularities and minor discrepancies between the root canal wall and core-filling material Expressed through lateral or accessory canals
* Can assist in microbial control
* Act as lubricant
* Can have adhesive property to dentin

The evolution of newer techniques, instruments, materials, and better understanding of canal anatomy, has changed the face of endodontics completely. One concept that has emerged is the single-visit root canal therapy. Single-visit root canal treatment (RCT) has become a common practice and offers several advantages, including a reduced flare-up rate, decreased number of operative procedures, and no risk of interappointment leakage through temporary restorations.

The major consideration regarding one-appointment endodontics has been the concern about postoperative pain . Various studies have evaluated the post-endodontic pain difference between single- and multiple-visit RCT, but most studies have ruled out any significant difference in postoperative pain .

It has been suggested that bioceramic materials improve the outcome of endodontic treatment by promoting the differentiation of odontoblasts and by releasing biologically active substances . The bioceramic materials have been shown to be less cytotoxic compared with resin-based AH Plus (Dentsply Maillefer, Ballaigues, Switzerland) in vitro . However, AH Plus (FKG Dentaire SA, La Chaux-de-Fonds, Switzerland) exhibited stronger bonding capacity and higher radiopacity compared with bioceramic sealers. The clinical significance of these characteristics is still unclear. Data on the clinical behavior of bioceramic sealers are scarce and of great interest.

ELIGIBILITY:
Inclusion Criteria:

* Permanent teeth with fully formed apex
* Teeth with vital pulp
* Teeth with no periapical radiolucency
* Patients having preoperative pain

Exclusion Criteria:

* Teeth with incompletely formed apex
* Teeth requiring secondary endodontic treatment
* Patients having complicating systemic disease such as diabetes, malignancy, pregnancy, central nervous system disorders, Cardiovascular system disorders, respiratory disorders, asthma patients, psychiatric disorders, immunocompromised patients,
* Patients taking anti-inflammatory or antibiotics
* Patients giving history of analgesic or antibiotic intake 1 week before treatment
* Patients below 18 years of age,
* Patients above 65 years of age
* Patients having history of peptic ulcer or gastrointestinal bleeding,
* Teeth having calcified canals,
* Teeth having multiple canals or multirooted teeth,
* Teeth affected with periodontal disease.
* Teeth tender on percussion,
* Teeth having procedural errors such as transportation, perforation, and missed canals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of postoperative pain | 6th hours
  Intensity of postoperative pain after using two types of sealers will be measured using a visual analog scale (VAS) after treatment
Intensity of postoperative pain | 12th hours
  Intensity of postoperative pain after using two types of sealers will be measured using a visual analog scale (VAS) after treatment
Intensity of postoperative pain | 24th hours
  Intensity of postoperative pain after using two types of sealers will be measured using a visual analog scale (VAS) after treatment

SECONDARY OUTCOMES:
intensity of postoperative pain | 48th hours
  Intensity of postoperative pain will be measured using a visual analog scale (VAS) after treatment
intensity of postoperative pain | 72nd hours
  Intensity of postoperative pain will be measured using a visual analog scale (VAS) after treatment
intensity of postoperative pain | 5th day
  Intensity of postoperative pain will be measured using a visual analog scale (VAS) after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hany Sadek, PHD, Study Director — Cairo University

REFERENCES:
- [Result] Graunaite I, Skucaite N, Lodiene G, Agentiene I, Machiulskiene V. Effect of Resin-based and Bioceramic Root Canal Sealers on Postoperative Pain: A Split-mouth Randomized Controlled Trial. J Endod. 2018 May;44(5):689-693. doi: 10.1016/j.joen.2018.02.010. Epub 2018 Mar 20. PMID 29571915
- [Result] Atav Ates A, Dumani A, Yoldas O, Unal I. Post-obturation pain following the use of carrier-based system with AH Plus or iRoot SP sealers: a randomized controlled clinical trial. Clin Oral Investig. 2019 Jul;23(7):3053-3061. doi: 10.1007/s00784-018-2721-6. Epub 2018 Nov 5. PMID 30397735